CLINICAL TRIAL: NCT04819100
Title: LIBRETTO-432: A Placebo-controlled Double-Blinded Randomized Phase 3 Study of Adjuvant Selpercatinib Following Definitive Locoregional Treatment in Participants With Stage IB-IIIA RET Fusion-Positive NSCLC
Brief Title: A Study of Selpercatinib After Surgery or Radiation in Participants With Non-Small Cell Lung Cancer (NSCLC)
Acronym: LIBRETTO-432
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Loxo Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18126; J2G-MC-JZJX (Other: Eli Lilly and Company); 2020-005191-35 (EudraCT Number); 2023-506784-33-00 (Other: EU Trial Number)
Record Dates: First submitted 2021-03-25; First posted 2021-03-26 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — selpercatinib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Selpercatinib (Experimental): Selpercatinib administered orally.
  Interventions: Drug: Selpercatinib
- Placebo (Placebo Comparator): Placebo administered orally.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Selpercatinib — Administered orally.
  Other Names: LY3527723; LOXO-292
  Arms: Selpercatinib
Drug: Placebo — Administered orally.
  Arms: Placebo

SUMMARY:
The reason for this study is to see if the study drug, selpercatinib, compared to placebo is effective and safe in delaying cancer return in participants with early-stage non-small cell lung cancer (NSCLC), who have already had surgery or radiation. Participants who are assigned to placebo and stop the study drug because their disease comes back or gets worse have the option to potentially crossover to selpercatinib. Participation could last up to three years.

ELIGIBILITY:
Inclusion Criteria:

* Must have histologically confirmed Stage IB, II, or IIIA NSCLC.
* Must have an activating RET gene fusion in tumor based on polymerase chain reaction (PCR), next generation sequencing (NGS), or another molecular test per sponsor's approval.
* Must have received definitive locoregional therapy with curative intent (surgery or radiotherapy) for Stage IB, II, or IIIA NSCLC.

  -- Must have undergone the available anti-cancer therapy (including chemotherapy or durvalumab) or not be suitable for it, based on the investigator's discretion.
* Maximum time allowed between definitive therapy completion and randomization must be:

  * 10 weeks if no chemotherapy was administered
  * 26 weeks if adjuvant chemotherapy was administered
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Adequate hematologic, hepatic, and renal function.
* Willingness of men and women of reproductive potential to observe conventional and highly effective birth control for the duration of the study and for at least 2 weeks after last dose of study drug.

Exclusion Criteria:

* Additional oncogenic drivers in NSCLC, if known.
* Evidence of small cell lung cancer.
* Clinical or radiologic evidence of disease recurrence or progression following definitive therapy.
* Known or suspected interstitial fibrosis or interstitial lung disease or history of (noninfectious) pneumonitis that required steroids.
* Clinically significant active cardiovascular disease or history of myocardial infarction within six months prior to planned start of selpercatinib or prolongation of the QT interval corrected for heart rate using Fridericia's formula (QTcF) greater than 470 milliseconds.
* Have known uncontrolled human immunodeficiency virus (HIV)-1/2 infection.
* Have known active hepatitis B or C.
* Active uncontrolled systemic bacterial, viral, or fungal infection or serious ongoing intercurrent illness, such as hypertension or diabetes, despite optimal treatment.
* Major surgery within 4 weeks prior to planned start of selpercatinib.
* Clinically significant active malabsorption syndrome or other condition likely to affect gastrointestinal absorption of the study drug.
* Other malignancy unless nonmelanoma skin cancer, carcinoma in situ of the cervix or other in situ cancers or a malignancy diagnosed greater than or equal to two years previously and not currently active.
* Pregnancy or lactation.
* Prior treatment with a selective RET inhibitor (e.g. selpercatinib or pralsetinib).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2021-12-20 (Actual); Primary Completion 2026-01-12 (Actual); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Event-Free Survival (EFS) | Randomization to disease recurrence/progression or death from any cause (estimated as up to 7 years)
  EFS by Investigator Assessment in the Primary Analysis Population

SECONDARY OUTCOMES:
EFS | Randomization to disease recurrence/progression or death from any cause (estimated as up to 7 years)
  EFS by investigator assessment in the overall population
Overall Survival (OS) | Randomization to death from any cause (estimated as up to 9 years)]
  OS
EFS | Randomization to disease recurrence/progression or death from any cause (estimated as up to 7 years)]
  EFS by blinded independent central review (BICR)
Time to Distant Disease Recurrence in the Central Nervous System (CNS) | Randomization to disease recurrence/progression or death from any cause (estimated as up to 7 years)
  Time to distant disease recurrence in the CNS by investigator assessment and BICR
Progression Free Survival on the Next Line of Treatment (PFS2) | Randomization to disease progression on the next line of treatment or death from any cause (estimated as up to 9 years)
  PFS2 by investigator assessment
Positive Predictive Value (PPV) of Rearranged during Transfection (RET) Tests from Investigator-Identified Laboratories with Respect to the Lilly-Designated RET Test | Baseline
  PPV of RET Tests from Investigator-Identified Laboratories with Respect to the Lilly-Designated RET Test
Mean Change from Baseline over Time in NSCLC Symptoms | Baseline to treatment discontinuation (estimated as up to 3 years)
  NSCLC symptoms will be measured using the 7-item NSCLC Symptom Assessment Questionnaire (NSCLC-SAQ). The NSCLC-SAQ measures the severity/frequency of the following core symptoms: Cough, pain, dyspnea, fatigue, and appetite. Raw scores range from 0 to 4 and the total score ranges from 0-20. Higher scores represent worse symptoms.
Mean Change from Baseline over Time in Physical Function | Baseline to treatment discontinuation (estimated as up to 3 years)
  Physical function will be measured by the 5 physical function items in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC-QLQ-C30) (also known as the EORTC IL 19 questionnaire). Raw scores range from 0-20. Higher scores indicate worst function.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (211):
- United States (15):
  - UCLA Hematology/Oncology - Santa Monica, Los Angeles, California
  - Stockton Hematology Oncology Group, Stockton, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - GenesisCare, Aventura, Florida
  - GenesisCare - Boca Raton, Boca Raton, Florida
  - USO-Cancer Care Center of Brevard, Inc., Palm Bay, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic in Rochester, Minnesota, Rochester, Minnesota
  - USO-New York Oncology Hematology, P.C, Latham, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - USO - Alliance Cancer Specialists, PC, Horsham, Pennsylvania
  - Sarah Cannon Research Institute SCRI, Nashville, Tennessee
  - Tennessee Oncology Nashville, Nashville, Tennessee
  - USO-Texas Oncology-Central/South Texas, Austin, Texas
  - US Oncology, The Woodlands, Texas
- Australia (8):
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Rockhampton Hospital, Rockhampton, Queensland
  - The Townsville Hospital, Townsville, Queensland
  - Ballarat Health Services, Ballarat Central, Victoria
  - Bendigo Health Care Group, Bendigo, Victoria
  - Goulburn Valley Health, Shepparton, Victoria
  - South West Healthcare, Warrnambool, Victoria
  - Border Medical Oncology, Wodonga, Victoria
- Austria (2):
  - Landeskrankenhaus Feldkirch, Feldkirch, Vorarlberg
  - Klinik Floridsdorf, Vienna
- Belgium (6):
  - Antwerp University Hospital, Edegem, Antwerpen
  - Cliniques universitaires Saint-Luc, Brussels, Bruxelles-Capitale, Région de
  - Université Catholique de Louvain-Namur - Centre Hospitalier Universitaire Dinant-Godinne - Site Godinne, Yvoir, Namur
  - Clinique Saint Pierre, Ottignies, Wallonne, Région
  - AZ Delta vzw, Roeselare, West-Vlaanderen
  - CHU UCL Namur/Site Sainte Elisabeth, Namur
- Brazil (12):
  - Nucleo de Oncologia da Bahia, Salvador, Estado de Bahia
  - Sirio-Libanes Brasilia - Centro de Oncologia - Asa Sul, Brasília, Federal District
  - Oncocentro de Minas Gerais, Belo Horizonte, Minas Gerais
  - Centro Oncológico do Triângulo, Uberlândia, Minas Gerais
  - Multihemo, Recife, Pernambuco
  - Hospital São Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Hospital BP, São Paulo, São Paulo
  - Instituto D'Or de Pesquisa e Ensino (IDOR), São Paulo, São Paulo
  - Instituto de Educação, Pesquisa e Gestão em Saúde, Rio de Janeiro
  - Centro Paulista de Oncologia Clínica, São Paulo
  - Núcleo de Pesquisa Clínica da Rede São Camilo, São Paulo
  - Sociedade Beneficente Israelita Brasileira Hospital Albert Einstein, São Paulo
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada
- China (19):
  - Beijing Friendship Hospital, Beijing, Beijing Municipality
  - Beijing Cancer hospital, Beijing, Beijing Municipality
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - Southern Medical University Nanfang Hospital, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Xiangya Hospital, Central South University, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jilin Cancer Hospital, Changchun, Jilin
  - Tangdu Hospital of Fourth Military Medical University of Chinese People's Liberation Army, Xi'an, Shaanxi
  - Jinan Central Hospital, Jinan, Shandong
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - the Third People's Hospital of Chengdu, Chengdu, Sichuan
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - First Affiliated Hosp of College of Med, Zhejiang University, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Tongji Medical College of Huazhong University of Science and Technology, Wuhan
- Czechia (3):
  - Masarykuv onkologicky ustav, Brno, Brno-město
  - Nemocnice AGEL Ostrava - Vitkovice a.s., Ostrava, Ostrava Město
  - Fakultni nemocnice Bulovka, Prague, Praha 8
- Odense Universitetshospital, Odense, Region Syddanmark, Denmark
- France (7):
  - Centre Leon Berard, Lyon, Auvergne-Rhône-Alpes
  - Assistance Publique Hôpitaux de Marseille - Hôpital de la Timone, Marseille, Bouches-du-Rhône
  - CHU Charles Nicolle, Rouen, Haute-Normandie
  - Centre Chirurgical Marie Lannelongue, Le Plessis-Robinson, Hauts-de-Seine
  - Hospices Civils de Lyon - Hopital Louis Pradel, Lyon, Rhône
  - Gustave Roussy, Villejuif, Val-de-Marne
  - Hopitaux Universitaires Paris Centre-Hopital Cochin, Paris
- Germany (12):
  - Thoraxklinik-Heidelberg gGmbH, Heidelberg, Baden-Wurttemberg
  - Klinik Löwenstein, Löwenstein, Baden-Wurttemberg
  - Asklepios Fachkliniken München-Gauting, Gauting, Bavaria
  - Klinikum der Ludwig-Maximilians-Universitaet Muenchen, München, Bavaria
  - Lungenfachklinik Immenhausen, Immenhausen, Hesse
  - Franziskus-Hospital Harderberg, Georgsmarienhütte, Lower Saxony
  - KRH, Klinikum Siloah, Hanover, Lower Saxony
  - Universitätsklinikum Münster - Albert Schweitzer Campus, Münster, North Rhine-Westphalia
  - LungenClinic Grosshansdorf, Großhansdorf, Schleswig-Holstein
  - Charite Universitätsmedizin Berlin Campus Benjamin Franklin, Berlin
  - Evangelische Lungenklinik Berlin, Berlin
  - Asklepios Klinik Harburg, Hamburg
- Greece (7):
  - University Hospital of Patras, Pátrai, Achaḯa
  - Agios Savvas Regional Cancer Hospital, Athens, Attikí
  - Errikos Dunant Hospital Center, Athens, Attikí
  - Sotiria Thoracic Diseases Hospital of Athens, Athens, Attikí
  - University General Hospital of Heraklion, Heraklion, Irakleío
  - European Interbalkan Medical Center, Thessaloniki, Thessaloníki
  - G. Papanikolaou General Hospital, Thessaloniki, Thessaloníki
- Hong Kong (3):
  - Hong Kong United Oncology Centre, Hong Kong
  - Princess Margaret Hospital, Lai Chi Kok
  - Queen Elizabeth Hospital, Yau Ma Tei
- India (5):
  - Regional Cancer Centre - Thiruvananthapuram, Thiruvananthapuram, Kerala
  - Tata Memorial Hospital, Mumbai, Maharashtra
  - Rashtrasant Tukdoji Regional Cancer Hospital, Nagpur, Maharashtra
  - HCG Manavata Cancer Centre, Nashik, Maharashtra
  - Rajiv Gandhi Cancer Institute And Research Centre, New Delhi, National Capital Territory of Delhi
- Israel (3):
  - Sheba Medical Center, Ramat Gan, Central District
  - Hadassah Medical Center, Jerusalem, Jerusalem
  - Rambam Health Care Campus, Haifa, Ḥeifā
- Italy (6):
  - Instituto Tumori Giovanni Paolo II, Bari, Apulia
  - ASST Grande Ospedale Metropolitano Niguarda, Milan, Milano
  - Humanitas, Rozzano, Milano
  - Azienda Ospedaliera Dei Colli, Naples, Napoli
  - Azienda Sanitaria Ospedaliera S Luigi Gonzaga, Orbassano, Torino
  - Istituto Oncologico Veneto IRCCS, Padua
- Japan (10):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Himeji Medical Center, Himeji, Hyōgo
  - Kanagawa cancer center, Yokohama, Kanagawa
  - Niigata Cancer Center Hospital, Niigata, Niigata
  - Shizuoka Cancer Center, Nakatogari, Shizuoka
  - Japanese Foundation for Cancer Research, Koto, Tokyo
  - Tottori University Hospital, Yonago, Tottori
  - Hiroshima University Hospital, Hiroshima
  - Osaka International Cancer Institute, Osaka
- Mexico (4):
  - Actualidad Basada en la Investigación del Cáncer, Guadalajara, Jalisco
  - Oncare Viaducto Napoles, Mexico City, Mexico City
  - Avix Investigación Clinica, S.C., Monterrey, Nuevo León
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey, Nuevo León
- Netherlands (2):
  - Ziekenhuis St. Jansdal, Harderwijk, Gelderland
  - Radboudumc, Nijmegen, Gelderland
- Oslo Universitetssykehus Ullevål, Oslo, Norway
- Krakowski Szpital Specjalistyczny im. Jana Pawa II, Krakow, Lesser Poland Voivodeship, Poland
- Pan American Center for Oncology Trials, Rio Piedras, Puerto Rico
- Institutul Oncologic, Cluj-Napoca, Romania
- Russia (4):
  - Arkhangelsk Clinical Oncological Dispensary, Arkhangelsk, Arkhangelskaya oblast
  - Hadassah Medical, Moscow, Moscow
  - First Pavlov State Medical University of Saint Petersburg, Saint Petersburg, Sankt-Peterburg
  - Scientific research institution of oncology named after N.N. Petrov, Saint Petersburg
- Singapore (2):
  - Parkway Cancer Centre - Gleneagles Hospital, Singapore, Central Singapore
  - Tan Tock Seng Hospital, Singapore, Central Singapore
- South Korea (10):
  - Chonnam National University Hwasun Hospital, Hwasun, Jeonranamdo
  - National Cancer Center, Goyang-si, Kyǒnggi-do
  - Seoul National University Bundang Hospital, Seongnam, Kyǒnggi-do
  - Pusan National University Hospital, Busan, Pusan-Kwangyǒkshi
  - Seoul National University Hospital, Seoul, Seoul-teukbyeolsi [Seoul]
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul-teukbyeolsi [Seoul]
  - Asan Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - Samsung Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - Korea University Guro Hospital, Seoul, Seoul-teukbyeolsi [Seoul]
  - Kyungpook National University Chilgok Hospital, Deagu, Taegu-Kwangyǒkshi
- Spain (27):
  - CHUS - Hospital Clinico Universitario, Santiago de Compostela, A Coruña [La Coruña]
  - Hospital Universitario Puerta del Mar, Cadiz, Andalusia
  - Hospital Universitario Reina Sofia, Córdoba, Andalusia
  - Institut Català d'Oncologia (ICO) - Badalona, Badalona, Barcelona [Barcelona]
  - Parc de Salut Mar - Hospital del Mar, Barcelona, Barcelona [Barcelona]
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [Barcelona]
  - Instituto Catalan de Oncologia - Hospital Duran i Reynals, L'Hospitalet Del Llobregat, Barcelona [Barcelona]
  - Hospital de Mataró, Mataró, Barcelona [Barcelona]
  - Complejo Asistencial Universitario de León - Hospital de León, León, Castille and León
  - Hospital Universitari Dexeusa, Barcelona, Catalunya [Cataluña]
  - Hospital Clínic de Barcelona, Barcelona, Catalunya [Cataluña]
  - Hospital Son Llàtzer, Palma, Illes Balears [Islas Baleares]
  - Hospital Lucus Augusti, Lugo, Lugo [Lugo]
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid, Comunidad de
  - Hospital Universitario 12 de Octubre, Madrid, Madrid, Comunidad de
  - Hospital Clínico Universitario Virgen de la Arrixaca, El Palmar, Murcia, Murcia, Región de
  - Complexo Hospitalario Universitario de Ourense, Ourense, Ourense [Orense]
  - CHUVI- Hospital Alvaro Cunqueiro, Pontevedra, Pontevedra [Pontevedra]
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Hospital Universitari Sant Joan de Reus, Reus, Tarragona [Tarragona]
  - Hospital General Universitario de Albacete, Albacete
  - MD Anderson Cancer Center, Madrid
  - Hospital Clinico San Carlos, Madrid
  - H.R.U Málaga - Hospital General, Málaga
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
- Sahlgrenska Universitetssjukhuset, Gothenburg, Västra Götalands Län [se-14], Sweden
- Taiwan (10):
  - Changhua Christian Hospital, Changhua County, Changhua
  - Chang Gung Memorial Hospital at Kaohsiung, Kaohsiung Niao Sung Dist, Kaohsiung
  - Chung Shan Medical University Hospital, Taichung, Taichung
  - Chi Mei Hospital - Liouying Branch, Tainan, Tainan
  - National Taiwan University Cancer Center (NTUCC), Taipei City, Taipei
  - Taipei Veterans General Hospital, Taipei City, Taipei
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District
- Turkey (Türkiye) (15):
  - Ege Universitesi Hastanesi, Bornova, İzmir
  - Izmir Medical Park Hospital, Izmir, Karsiyaka, İzmir
  - Baskent University Dr. Turgut Noyan Research and Training Center, Adana
  - Adana City Hospital, Adana
  - Abdurrahman Yurtaslan Ankara Oncology, education and Research Hospital, Ankara
  - Ankara Bilkent Şehir Hastanesi, Ankara
  - Memorial Antalya Hospital, Antalya
  - Uludag Universitesi, Bursa
  - Dicle Üniversitesi, Diyarbakır
  - Trakya University, Edirne
  - Medipol Mega Universite Hastanesi, Istanbul
  - Acıbadem Maslak Hastanesi, Istanbul
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi, Istanbul
  - Izmir Katip Celebi Ataturk Egitim Arastirma Hastanesi, Izmir
  - İnönü Üniversitesi Turgut Özal Tıp Merkezi Eğitim ve Araştırma Hastanesi, Malatya
- Ukraine (7):
  - Medical Center "Mriya Med-Service", Kryvyi Rih, Dnipropetrovsk Oblast
  - CNPE "Regional Center of Oncology", Kharkiv, Kharkivs’ka Oblast’
  - Municipal non-profit enterprise'Odesa Regional Clinical Hospital'of Odesa Regional Council, Odesa, Odesa Oblast
  - Sumy regional clinical oncological dispensary, Sumy, Sumska Oblast
  - Communal Noncommercial Enterprise "Podillia Regional Oncology Center Of Vinnytsia Regional Council", Vinnytsia, Vinnytsia Oblast
  - "Oncolife" LLC, Zaporizhzhia, Zaporizhzhia Oblast
  - Municipal non-profit enterprise "Kyiv City Clinical Oncology Center" of executive body of Kyiv City Counci -T, Kyiv
- United Kingdom (5):
  - Chelsea and Westminster Hospital NHS Foundation Trust, London, England
  - Royal Brompton Hospital, London, Kensington and Chelsea
  - University College London Hospital, London, London, City of
  - City Hospital, Nottingham University Hospitals, Nottingham
  - New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Tsuboi M, Goldman JW, Wu YL, Johnson ML, Paz-Ares L, Yang JC, Besse B, Su W, Chao BH, Drilon A. LIBRETTO-432, a phase III study of adjuvant selpercatinib or placebo in stage IB-IIIA RET fusion-positive non-small-cell lung cancer. Future Oncol. 2022 Sep;18(28):3133-3141. doi: 10.2217/fon-2022-0656. Epub 2022 Aug 11. PMID 35950566
- See also: A Study of Selpercatinib After Surgery or Radiation in Participants With Non-Small Cell Lung Cancer (NSCLC) (LIBRETTO-432) — https://trials.lilly.com/ext/trial?id=J2G-MC-JZJX